CLINICAL TRIAL: NCT02408016
Title: Phase I/II Study in WT1-Expressing Non-small Cell Lung Cancer and Mesothelioma, Comparing Cellular Adoptive Immunotherapy With Polyclonal Autologous Central Memory to Naïve CD8+ T Cells That Have Been Transduced to Express a WT1-Specific T-Cell Receptor
Brief Title: Genetically Modified T Cells in Treating Patients With Stage III-IV Non-small Cell Lung Cancer or Mesothelioma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Terminated due to loss of funding
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Aude Chapuis, Associate Professor, Fred Hutchinson Cancer Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2727.00; NCI-2015-00329 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2727; 2727.00 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2015-03-31; First posted 2015-04-03 (Estimated); Results first posted 2021-09-13 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-08

CONDITIONS: Advanced Pleural Malignant Mesothelioma; HLA-A*0201 Positive Cells Present; Recurrent Non-Small Cell Lung Carcinoma; Recurrent Pleural Malignant Mesothelioma; Stage III Non-Small Cell Lung Cancer AJCC v7; Stage III Pleural Malignant Mesothelioma AJCC v7; Stage IIIA Non-Small Cell Lung Cancer AJCC v7; Stage IIIB Non-Small Cell Lung Cancer AJCC v7; Stage IV Non-Small Cell Lung Cancer AJCC v7; Stage IV Pleural Malignant Mesothelioma AJCC v7; WT1 Positive
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Mesothelioma, Malignant | interventions — aldesleukin; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm I, Stage I (T lymphocytes, cyclophosphamide, IL-2) (Experimental): Patients receive autologous WT1-TCRc4 gene-transduced CD8-positive Tcm/Tn lymphocytes IV on days 0 and 14, cyclophosphamide IV on days 11 and 12, and aldesleukin SC BID for 14 days. Patients who have received radiation to the chest/lung tissue may receive gene-transduced T lymphocytes 90 days after completion of radiation.
  Interventions: Biological: Aldesleukin; Biological: Autologous WT1-TCRc4 Gene-transduced CD8-positive Tcm/Tn Lymphocytes; Drug: Cyclophosphamide; Other: Laboratory Biomarker Analysis
- Arm I, Stage II (T lymphocytes, cyclophosphamide, IL-2) (Experimental): Patients receive cyclophosphamide IV on days -3 and -2, autologous WT1-TCRc4 gene-transduced CD8-positive Tcm/Tn lymphocytes IV on day 0, and aldesleukin SC BID for 14 days.
  Interventions: Biological: Aldesleukin; Biological: Autologous WT1-TCRc4 Gene-transduced CD8-positive Tcm/Tn Lymphocytes; Drug: Cyclophosphamide; Other: Laboratory Biomarker Analysis
- Arm II (T lymphocytes, IL-2, surgery) (Experimental): Patients receive autologous WT1-TCRc4 gene-transduced CD8-positive Tcm/Tn lymphocytes IV between 24-96 hours after the last dose of chemotherapy and receive aldesleukin SC BID for 14 days. Patients then undergo surgery within 3-4 weeks after the T-cell infusion.
  Interventions: Biological: Aldesleukin; Biological: Autologous WT1-TCRc4 Gene-transduced CD8-positive Tcm/Tn Lymphocytes; Other: Laboratory Biomarker Analysis; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Biological: Aldesleukin — Given SC
  Other Names: 125-L-Serine-2-133-interleukin 2; Proleukin; r-serHuIL-2; Recombinant Human IL-2; Recombinant Human Interleukin-2
Biological: Autologous WT1-TCRc4 Gene-transduced CD8-positive Tcm/Tn Lymphocytes — Given IV
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
  Arms: Arm I, Stage I (T lymphocytes, cyclophosphamide, IL-2); Arm I, Stage II (T lymphocytes, cyclophosphamide, IL-2)
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Therapeutic Conventional Surgery — Undergo surgical resection
  Arms: Arm II (T lymphocytes, IL-2, surgery)

SUMMARY:
This phase I/II trial studies the side effects and best dose of genetically modified T cells in treating patients with stage III-IV non-small cell lung cancer (NSCLC) or mesothelioma. Many types of cancer cells, including NSCLC and mesothelioma, but not most normal cells, have a protein called Wilms tumor (WT)1 on their surfaces. This study takes a type of immune cell from patients, called T cells, and modifies their genes in the laboratory so that they are programmed to find cells with WT1 and kill them. The T cells are then given back to the patient. Cyclophosphamide and aldesleukin may also stimulate the immune system to attack cancer cells. Giving cyclophosphamide and aldesleukin with laboratory-treated T cells may help the body build an immune response to kill tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the safety, and potential toxicities associated with treating patients with metastatic NSCLC and mesothelioma with polyclonal autologous central memory and naive cluster of differentiation (CD)8+ T cells that have been transduced to express a WT1-specific T-cell receptor (TCR) (Arm 1 and Arm 2).

II. Determine the feasibility of treating patients with metastatic NSCLC and mesothelioma with polyclonal autologous central memory and naive CD8+ T cells that have been transduced to express a WT1-specific TCR (Arm 1 and Arm 2).

III. Determine and compare the in vivo persistence in blood and tumor of transferred polyclonal autologous central memory and naive CD8+ T cells that have been transduced to express a WT1-specific TCR (Arm 1 and Arm 2).

EXPLORATORY OBJECTIVES:

I. Determine the antitumor efficacy for patients with metastatic NSCLC and mesothelioma (Arm 1), as measured by time to progression (TTP) based on the Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria.

II. Determine the in vivo functional capacity of adoptively transferred polyclonal autologous CD8+ T cells that have been transduced to express a WT1-specific TCR, and assess the acquisition of phenotypic characteristics associated with T cell exhaustion (Arm 1 and Arm 2).

III. Determine the migration to tumor sites of adoptively transferred polyclonal autologous CD8+ T cells that have been transduced to express a WT1-specific TCR (Arm 2).

IV. Evaluate the tumor response and T cell infiltration in tumors of patients with stage IIIA NSCLC treated in the neo-adjuvant setting.

OUTLINE: This is a phase I, dose-escalation study of autologous WT1-TCRc4 gene-transduced CD8-positive Tcm/Tn lymphocytes followed by a phase II study. Patients are assigned to 1 of 3 treatment arms.

ARM I, STAGE I: Patients receive autologous WT1-TCRc4 gene-transduced CD8-positive Tcm/Tn lymphocytes intravenously (IV) on days 0 and 14, cyclophosphamide IV on days 11 and 12, and aldesleukin (IL-2) subcutaneously (SC) twice daily (BID) for 14 days. Patients who have received radiation to the chest/lung tissue may receive T lymphocytes 90 days after completion of radiation.

ARM I, STAGE II: Patients receive cyclophosphamide IV on days -3 and -2, autologous WT1-TCRc4 gene-transduced CD8-positive Tcm/Tn lymphocytes IV on day 0, and aldesleukin SC BID for 14 days.

ARM II: Patients receive autologous WT1-TCRc4 gene-transduced CD8-positive Tcm/Tn lymphocytes IV between 24-96 hours after the last dose of chemotherapy and receive aldesleukin SC BID for 14 days. Patients then undergo surgery within 3-4 weeks after the T-cell infusion.

After completion of study treatment, patients are followed up at 3, 6, and 12 months and then annually for 14 years.

ELIGIBILITY:
Inclusion Criteria:

* ELIGIBILITY FOR ENROLLMENT/SCREENING (ARMS 1 AND 2): Histopathological documentation of NSCLC or mesothelioma
* ELIGIBILITY FOR ENROLLMENT/SCREENING (ARMS 1 AND 2): Patients must be able to give informed consent
* ELIGIBILITY FOR ENROLLMENT/SCREENING (ARMS 1 AND 2): Patients must be able to provide blood and tumor samples and undergo the procedures required for this protocol
* Arm 2 ONLY: Surgically operable NSCLC or mesothelioma
* ELIGIBILITY FOR TREATMENT ON ARM 1: Patients must express human leukocyte antigen (HLA)-A*0201
* ELIGIBILITY FOR TREATMENT ON ARM 1: Evidence of WT1 tumor expression
* ELIGIBILITY FOR TREATMENT ON ARM 1: Patients must have received at least one line of therapy for NSCLC or mesothelioma or previously documented to have declined therapy
* ELIGIBILITY FOR TREATMENT ON ARM 1: NSCLC patients with a mutation in epidermal growth factor receptor (EGFR) or anaplastic lymphoma kinase (ALK) must have demonstrated progression or intolerance to at least one of the corresponding targeted therapies (for example erlotinib or crizotinib)
* ELIGIBILITY FOR TREATMENT ON ARM 1: Bi-dimensionally measurable disease by palpation, clinical exam, or radiographic imaging (X-ray, computed tomography [CT] scan, positron emission tomography [PET] scan, magnetic resonance imaging [MRI], or ultrasound)
* ELIGIBILITY FOR TREATMENT ON ARM 1: Ninety days must have passed since the last doses of radiation or chemoradiation treatment involving lung tissue or thorax prior to T cell infusion (to avoid confounding pneumonitis)
* ELIGIBILITY FOR TREATMENT ON ARM 1: Patients treated with prior immunotherapy including and not limited to vaccines, cytokines, T cell stimulating agents, cytotoxic T lymphocyte antigen 4 (CTLA4) inhibitors and programmed death (PD)-1 check point inhibitors are allowed on therapy provided they did not have any severe grade 4 toxicities due to prior therapy and any toxicities due to prior therapy should have resolved, if resolvable to less than or equal to grade 1
* ELIGIBILITY FOR TREATMENT ON ARM 2: Patients must express HLA-A*0201
* ELIGIBILITY FOR TREATMENT ON ARM 2: Evidence of WT1 tumor expression
* ELIGIBILITY FOR TREATMENT ON ARM 2: Ninety days must have passed since the last definitive doses of radiation or chemoradiation treatment prior to T cell infusion (to avoid confounding pneumonitis)

Exclusion Criteria:

* EXCLUSION FOR ENROLLMENT/SCREENING (ARMS 1 AND 2)
* Eastern Cooperative Oncology Group (ECOG) performance status >= 2
* Active autoimmune disease (e.g., systemic lupus erythematosus, vasculitis, infiltrating lung disease, inflammatory bowel disease) in which possible progression during treatment would be considered unacceptable by the investigators
* Any condition or organ toxicity deemed by the principal investigator (PI) or the attending physician to place the patient at unacceptable risk for treatment on the protocol
* Men or women of reproductive ability who are unwilling to use effective contraception or abstinence; women of childbearing potential must have a negative urine pregnancy test within 2 weeks prior to first infusion
* Pregnant women and nursing mothers will be eligible for screening only to test HLA type by saliva or buccal swab and WT1 expression from previously collected tissue sample
* Clinically significant and ongoing immune suppression including, but not limited to, systemic immunosuppressive agents such as cyclosporine or corticosteroids, chronic lymphocytic leukemia (CLL), uncontrolled human immunodeficiency virus (HIV) infection, or solid organ transplantation
* EXCLUSION FOR TREATMENT (ARMS 1 AND 2)
* Exclusions for the leukapheresis procedure (this can be performed at a later time of symptoms resolve):

  * Infection, with or without antibiotic treatment
  * Recent hepatitis exposure (hepatitis B or C antigenemia)
  * Pregnancy or nursing
  * HIV or human T-lymphotropic virus (HTLV) infection
  * Positive result on standard test for syphilis (STS)
* Unable to generate antigen-specific WT1-specific CD8+ T cells for infusions; however, the patient will have the option to receive WT1-specific T-cells if a lower than planned number of cells is available
* Documented infections or known oral temperature > 38.2 degrees Celsius (C) fewer than 72 hours prior to receiving study treatment or systemic infection requiring chronic maintenance; the start of treatment may be delayed
* Systemic steroids should be stopped 2 weeks before the start of treatment; topical and inhaled steroids are allowed
* Untreated central nervous system (CNS) metastasis that are > 1 cm or symptomatic are not allowed; (patients with CNS metastases > 1 cm or symptomatic that have been treated and demonstrated to be radiologically and clinically stable for at least 4 weeks are allowed)
* White blood cells (WBC) < 2,000/ul
* Hemoglobin (Hb) < 8 g/dL
* Absolute neutrophil count (ANC) < 1,000/ul
* Platelets < 50,000/ul
* New York Heart Association functional class III-IV heart failure, symptomatic pericardial effusion, stable or unstable angina, symptoms of coronary artery disease (CAD), congestive heart failure, clinically significant hypotension or history of an ejection fraction of =< 30% (echocardiogram or multi-gated acquisition scan [MUGA])
* Clinically significant pulmonary dysfunction, as determined by medical history and physical exam; patients so identified will undergo pulmonary functions testing and those with forced expiratory volume in 1 second (FEV1) < 2.0 L or diffusion capacity of the lungs for carbon monoxide (DLCO) (corrected for Hb) < 50% will be excluded
* Creatinine > 1.5 x the upper limit of normal
* Aspartate aminotransferase/alanine aminotransferase (AST/ALT) > 5 x upper limits of normal (ULN)
* Bilirubin > 3 x ULN that cannot be attributed to NSCLC metastasis
* HIV or HTLV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-05-22 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia Lee, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 11 participants were enrolled, but only 10 participants were assigned to an arm/group.
Period: Overall Study
Arm/Group | Arm I, Stage I (T Lymphocytes, Cyclophosphamide, IL-2) | Arm I, Stage II (T Lymphocytes, Cyclophosphamide, IL-2) | Arm II (T Lymphocytes, IL-2, Surgery)
Started | 6 | 4 | 0
Completed | 0 | 1 | 0
Not Completed | 6 | 3 | 0
Not completed — Death | 6 | 1 | 0
Not completed — Physician Decision | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: No patients were treated in Arm II
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I, Stage I (T Lymphocytes, Cyclophosphamide, IL-2) | Arm I, Stage II (T Lymphocytes, Cyclophosphamide, IL-2) | Arm II (T Lymphocytes, IL-2, Surgery) | Total
Number analyzed (Participants) | 6 | 4 | 0 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 |  | 0
  Between 18 and 65 years | 4 | 0 |  | 4
  >=65 years | 2 | 4 |  | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 |  | 6
  Male | 2 | 2 |  | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 |  | 0
  Not Hispanic or Latino | 6 | 4 |  | 10
  Unknown or Not Reported | 0 | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 |  | 0
  Asian | 0 | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  | 0
  Black or African American | 0 | 0 |  | 0
  White | 6 | 4 |  | 10
  More than one race | 0 | 0 |  | 0
  Unknown or Not Reported | 0 | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 4 |  | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Based on the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0.
Time Frame: Up to 6 months after the first T cell infusion
Population: No patients were treated in Arm II.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I, Stage I (T Lymphocytes, Cyclophosphamide, IL-2) | Arm I, Stage II (T Lymphocytes, Cyclophosphamide, IL-2) | Arm II (T Lymphocytes, IL-2, Surgery)
Number analyzed (Participants) | 6 | 4 | 0
Participants | 6 | 3 | 0

2. Primary Outcome: Count of Patients for Which T Cells Are Successfully Generated and Infused and Whether Only TN or TCM Could be Generated
Description: There were products generated for 11 participants and 10 participants were treated on the study. 8 participants received an infusion with Tn and Tcm cells. 1 participant received infusions with only Tn cells. 1 participant received their last infusion with only Tcm cells. The one participant that was not treated did successfully have Tn and Tcm cells generated but they were not treated due to their condition worsening.
Time Frame: Up to 4 weeks
Population: No patients were treated in Arm II.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I, Stage I (T Lymphocytes, Cyclophosphamide, IL-2) | Arm I, Stage II (T Lymphocytes, Cyclophosphamide, IL-2) | Arm II (T Lymphocytes, IL-2, Surgery)
Number analyzed (Participants) | 6 | 4 | 0
Participants | 4 | 4 | 0

3. Primary Outcome: Persistence of Transduced T Cells
Description: In vivo persistence of cells generated from the TN subset with cells generated from the TCM subset will be directly compared within each patient by high throughput T-cell receptor (TCR) beta sequencing. The one-sample T test will be used to assess the difference in mean persistence between groups, in which the outcome for each patient is the time to disappearance of infused cytotoxic T lymphocytes.
Time Frame: Up to 100 days after the last T cell infusion
Population: No patients were treated in Arm II
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I, Stage I (T Lymphocytes, Cyclophosphamide, IL-2) | Arm I, Stage II (T Lymphocytes, Cyclophosphamide, IL-2) | Arm II (T Lymphocytes, IL-2, Surgery)
Number analyzed (Participants) | 6 | 4 | 0
Participants | NA — This outcome could not be assessed. Although we detected persistence if T cells by tetramer staining in all patients, the transduced cells came from the endogenous repertoire from each patient. As the pre-T cell infusion leaves were elevated, we could not detect changes in TN vs TCM using high-throughput TCR sequencing. | NA — This outcome could not be assessed. Although we detected persistence if T cells by tetramer staining in all patients, the transduced cells came from the endogenous repertoire from each patient. As the pre-T cell infusion leaves were elevated, we could not detect changes in TN vs TCM using high-throughput TCR sequencing. | 0

4. Other Pre Specified Outcome: Frequency of Transferred T Cells at Biopsied Tumor Sites Between the T Cell (Tn) and Memory T Cell (Tcm) Groups
Description: Frequency of transferred T cells at biopsied tumor sites between the Tn and Tcm groups will be assessed.
Time Frame: Up to 15 years
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Functional Capacity of Transferred Cells, Measured by Production of Intracellular Cytokines
Description: Tetramer+ cells from peripheral blood, if detectable and available in sufficient number, evaluated for production of intracellular cytokines including interferon-gamma (IFN-gamma), tumor necrosis factor alpha (TNF-alpha), and IL-2. Intranuclear Ki-67 expression assessed on recovered tetramer+ T cells. Based on available numbers, ex vivo proliferative capacity after infusion assessed by labeling cells with carboxyfluorescein succinimidyl ester dye and measuring dilution in response to peptide stimulation. Phenotype of tetramer+ antigen-specific cells assessed using established immunophenotyping
Time Frame: Up to 15 years
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Time to Progression (TTP) Based on Response Evaluation Criteria in Solid Tumors (RECIST) Criteria and RECIST 1.1 Mesothelioma Modified
Description: The potential efficacy of the infused cells will be assessed and the substrate cell (TN or TCM) that is most effective based on the TTP of patients who have persisting TN cells to that of patients who have persisting TCM cells 3 months after the last infusion will be determined.
Time Frame: 3 months after last infusion
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 12 months
Description: No patients were treated in Arm II.
Arm/Group | Arm I, Stage I (T Lymphocytes, Cyclophosphamide, IL-2) | Arm I, Stage II (T Lymphocytes, Cyclophosphamide, IL-2) | Arm II (T Lymphocytes, IL-2, Surgery)
All-Cause Mortality (participants affected / at risk) | 6/6 | 2/4 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/4 | 0/0
Other Adverse Events (participants affected / at risk) | 6/6 | 3/4 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I, Stage I (T Lymphocytes, Cyclophosphamide, IL-2) (N=6) | Arm I, Stage II (T Lymphocytes, Cyclophosphamide, IL-2) (N=4) | Arm II (T Lymphocytes, IL-2, Surgery) (N=0)
Fever (General disorders) | 2 (2) | 0 (0) | NA
Lymphocyte count decreased (Investigations) | 6 (9) | 3 (3) | NA
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | NA
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | NA
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | NA
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | NA
Fatigue (General disorders) | 0 (0) | 1 (2) | NA
White blood cell count decreased (Investigations) | 0 (0) | 1 (1) | NA
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-11): https://cdn.clinicaltrials.gov/large-docs/16/NCT02408016/Prot_SAP_000.pdf